CLINICAL TRIAL: NCT04272541
Title: Effectiveness of a Psychoeducation Program on Metabolic Syndrome, Cardiovascular Risk, Independency and Psychopatology in Patients With Severe Mental Illness
Brief Title: Effectiveness of a Psychoeducation Program in Patients With Severe Mental Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, José Manuel Pérez Mármol, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCT04272541
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Mental Health Disorder; Healthy Lifestyle
Keywords: cardiovascular risk; metabolic syndrome; independency; psychopathology
MeSH Terms: conditions — Mental Disorders; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation program (Active Comparator): The intervention program consists of psychopharmacology (standard intervention in mental health services) + individual psychoeducation (individual treatment including learning of Healthy Lifestyle). This program is implemented for three months, allocated in several sessions.
  Interventions: Behavioral: Psychoeducation program
- Habitual intervention (Active Comparator): Intervention program consists of psychopharmacology (standard intervention in mental health services). This program is implemented for three months.
  Interventions: Drug: Psychopharmacology intervention

INTERVENTIONS:
Behavioral: Psychoeducation program — Intervention program consisted of psychopharmacology + psychoeducation. This will be executed during 3 months, distribuited in several sessions.
  Other Names: Mixed treatment program
  Arms: Psychoeducation program
Drug: Psychopharmacology intervention — Intervention program consisted of psychopharmacology. This will be executed during 3 months.
  Other Names: Standard intervention
  Arms: Habitual intervention

SUMMARY:
Patients with Severe Mental Disorder (SMD) show a life expectancy of 13 to 30 years lower than the general population. Among the factors that determine this expectancy are cardiovascular risk and the metabolic syndrome. The objective of the present study will be to evaluate the effectiveness of a rehabilitative intervention comprinsing a psychopharmacology and psychoeducation program on cardiovascular risk, metabolic syndrome, independency for activities of daily living and psychopathological symptoms.

DETAILED DESCRIPTION:
It will be selected sixty patients diagnosed with SMD from a community Mental Health Unit from Spain. It will be implemented a intervention program consisted of psychopharmacology + psychoeducation on healthy living habits during three months. The patients will be evaluated at the beginning, at three months and at six months follow-up for weight, waist circumference, waist-hip ratio, body mass index, cardiovascular risk, independency and psychopathology.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years old,
* A body mass index higher than 30
* Psychopathologically stabilized

Exclusion Criteria:

* Cognitive impairment

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
weight | Change from Baseline in weight at 3 and 6 months
  This measurement registers weight in Kg

SECONDARY OUTCOMES:
waist circumference | Change from Baseline in waist circumference at 3 and 6 months
  This measurement registers waist circumference in cm
waist-hip ratio | Change from Baseline in waist-hip ratio at 3 and 6 months
  Waist-hip ratio will be calculated
Framingham scale | Change from Baseline in Framingham scale at 3 and 6 months
  The Framingham Risk Score is a gender-specific algorithm used to estimate the 10-year cardiovascular risk of an individual.
Global Assesment of funtioning Scale | Change from Baseline in Global Assesment of funtioning Scale at 3 and 6 months
  This scale evaluates psychological, social, and occupational functioning dimensions on a hypothetical continuum of mental health-illness.
PANNS | Change from Baseline in PANNS at 3 and 6 months
  The Positive and Negative Syndrome Scale for mental disorder

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Pérez Mármol, PhD, Principal Investigator — Department of Physiotherapy. Faculty of Health Sciences, University of Granada
Locations (1):
- José Manuel Pérez Mármol, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No